CLINICAL TRIAL: NCT02980133
Title: A 12-Week, Randomized, Double-Blind, Placebo-Controlled, Efficacy and Safety Study of Fluticasone Propionate Multidose Dry Powder Inhaler Compared With Fluticasone Propionate/Salmeterol Multidose Dry Powder Inhaler in Patients Aged 4 Through 11 Years With Persistent Asthma
Brief Title: Study of Fluticasone Propionate Multidose Dry Powder Inhaler Compared With Fluticasone Propionate/Salmeterol Multidose Dry Powder Inhaler
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FSS-AS-30003; 2016-003835-39 (EudraCT Number)
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo MDPI (Placebo Comparator): Participants received matching placebo via multidose dry powder inhaler (MDPI) for 12 weeks.
  Interventions: Drug: Placebo MDPI
- Fp MDPI 25 mcg BID (Experimental): Participants received 1 inhalation of 25 mcg fluticasone propionate (Fp) via MDPI twice daily (BID) (total daily dose: 50 mcg) for 12 weeks.
  Interventions: Drug: Fluticasone Propionate
- Fp MDPI 50 mcg BID (Experimental): Participants received 1 inhalation of 50 mcg fluticasone propionate via MDPI BID (total daily dose: 100 mcg) for 12 weeks.
  Interventions: Drug: Fluticasone Propionate
- FS MDPI 50/12.5 mcg BID (Experimental): Participants received 1 inhalation of 50/12.5 mcg fluticasone propionate/salmeterol (FS) via MDPI BID (total daily dose: 100/25 mcg) for 12 weeks.
  Interventions: Drug: Fluticasone Propionate/Salmeterol

INTERVENTIONS:
Drug: Fluticasone Propionate — Fluticasone propionate was administered via MDPI per the dose and schedule specified in the arm.
  Arms: Fp MDPI 25 mcg BID; Fp MDPI 50 mcg BID
Drug: Fluticasone Propionate/Salmeterol — Fluticasone propionate/salmeterol was administered via MDPI per the dose and schedule specified in the arm.
  Arms: FS MDPI 50/12.5 mcg BID
Drug: Placebo MDPI — Matching placebo was administered via MDPI per the schedule specified in the arm.
  Arms: Placebo MDPI

SUMMARY:
This study is to evaluate the safety and efficacy of fluticasone propionate and fluticasone propionate salmeterol in pediatric participants with a documented history of persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a diagnosis of asthma as defined by the National Institutes of Health (NIH).
* The participant has persistent asthma with a FEV1 ≥50% and ≤90% of the value predicted for age, height, sex, and race at the screening visit (SV).
* The participant's persistent asthma is stable and is currently being treated with stable asthma therapy for at least 30 days before the SV. Participants currently on a short-acting β2-agonist (SABA) only, regimen or as needed (PRN), are not eligible.
* The participant has demonstrated ≥10% response to a bronchodilator from screening FEV1 within 30 minutes after 2 to 4 inhalations of albuterol/salbutamol.
* The participant (with assistance from parents/legal guardians/caregivers, as needed) is able to perform technically acceptable lung function assessments by handheld device.
* All participants must be able to replace their current SABA with albuterol/salbutamol hydrofluoroalkane (HFA) metered-dose inhaler (MDI) inhalation aerosol at the SV for use as needed for the duration of the study.

  * Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* The participant has a history of life-threatening asthma exacerbation that is defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest, or hypoxic seizures.
* The participant is pregnant or lactating or plans to become pregnant during the study period or within 30 days after the participant's last study-related visit.
* The participant has a known hypersensitivity to any corticosteroid, salmeterol, or any of the excipients in the investigational medicinal product (IMP) or rescue medication formulation (that is, lactose).
* The participant has been treated with any known strong cytochrome P450 (CYP) 3A4 inhibitors (for example, ketoconazole, ritonavir, clarithromycin) within 30 days before the SV or plans to be treated with any strong CYP3A4 inhibitor during the study.
* The participant currently smokes or has a smoking history. The participant must not have used tobacco products within the past year (for example, cigarettes, cigars, chewing tobacco, or pipe tobacco).
* The participant has had an asthma exacerbation requiring systemic corticosteroids within 30 days before the SV or has had any hospitalization for asthma within 2 months before the SV.
* The participant has used immunosuppressive medications within 30 days before the SV.
* The participant has untreated oral candidiasis at the SV. Participants with clinical visual evidence of oral candidiasis who agree to receive treatment and comply with appropriate medical monitoring may enter the run-in period.
* The participant has a history of a positive test for human immunodeficiency virus, active hepatitis B virus, or hepatitis C infection.
* The participant is an immediate relative of an employee of the clinical investigational center.
* A member of the participant's household is participating in the study at the same time.
* Vulnerable participants (that is, people kept in detention) are excluded from participation.

  * Additional criteria apply, please contact the investigator for more information

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 841 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2019-04-07 (Actual); Study Completion 2019-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (118):
- United States (77):
  - Teva Investigational Site 13881, Birmingham, Alabama
  - Teva Investigational Site 13883, Little Rock, Arkansas
  - Teva Investigational Site 13906, Bakersfield, California
  - Teva Investigational Site 14615, Corona, California
  - Teva Investigational Site 13892, Downey, California
  - Teva Investigational Site 13875, Fountain Valley, California
  - Teva Investigational Site 13904, Huntington Beach, California
  - Teva Investigational Site 13877, Huntington Beach, California
  - Teva Investigational Site 14668, Long Beach, California
  - Teva Investigational Site 13914, Napa, California
  - Teva Investigational Site 13918, Paramount, California
  - Teva Investigational Site 14618, Rolling Hills Estates, California
  - Teva Investigational Site 13912, Roseville, California
  - Teva Investigational Site 13847, Stockton, California
  - Teva Investigational Site 13848, Thousand Oaks, California
  - Teva Investigational Site 13856, Centennial, Colorado
  - Teva Investigational Site 13910, Colorado Springs, Colorado
  - Teva Investigational Site 13868, Longmont, Colorado
  - Teva Investigational Site 13913, Chiefland, Florida
  - Teva Investigational Site 14616, DeLand, Florida
  - Teva Investigational Site 13909, Homestead, Florida
  - Teva Investigational Site 13857, Loxahatchee Groves, Florida
  - Teva Investigational Site 13872, Miami, Florida
  - Teva Investigational Site 13907, Miami, Florida
  - Teva Investigational Site 13893, Miami, Florida
  - Teva Investigational Site 13886, Miami, Florida
  - Teva Investigational Site 13899, Miami, Florida
  - Teva Investigational Site 13864, Miami, Florida
  - Teva Investigational Site 13880, Miami, Florida
  - Teva Investigational Site 13870, Miami Lakes, Florida
  - Teva Investigational Site 14617, Miami Lakes, Florida
  - Teva Investigational Site 13916, Miami Springs, Florida
  - Teva Investigational Site 13911, Ocala, Florida
  - Teva Investigational Site 13876, Palmetto Bay, Florida
  - Teva Investigational Site 13844, Winter Park, Florida
  - Teva Investigational Site 13866, Gainesville, Georgia
  - Teva Investigational Site 13858, Savannah, Georgia
  - Teva Investigational Site 13896, Eagle, Idaho
  - Teva Investigational Site 13903, Idaho Falls, Idaho
  - Teva Investigational Site 13882, Springfield, Illinois
  - Teva Investigational Site 13887, Overland Park, Kansas
  - Teva Investigational Site 13851, Owensboro, Kentucky
  - Teva Investigational Site 13849, Rockville, Maryland
  - Teva Investigational Site 13865, Columbia, Missouri
  - Teva Investigational Site 13885, Columbia, Missouri
  - Teva Investigational Site 13891, Missoula, Montana
  - Teva Investigational Site 13897, Ocean City, New Jersey
  - Teva Investigational Site 13854, Verona, New Jersey
  - Teva Investigational Site 13908, Watertown, New York
  - Teva Investigational Site 13890, Charlotte, North Carolina
  - Teva Investigational Site 13863, Raleigh, North Carolina
  - Teva Investigational Site 13855, Canton, Ohio
  - Teva Investigational Site 13905, Milford, Ohio
  - Teva Investigational Site 13852, Oklahoma City, Oklahoma
  - Teva Investigational Site 13879, Oklahoma City, Oklahoma
  - Teva Investigational Site 13884, Oklahoma City, Oklahoma
  - Teva Investigational Site 13860, Tulsa, Oklahoma
  - Teva Investigational Site 13894, Tulsa, Oklahoma
  - Teva Investigational Site 13861, Medford, Oregon
  - Teva Investigational Site 13874, Pittsburgh, Pennsylvania
  - Teva Investigational Site 13895, Scottdale, Pennsylvania
  - Teva Investigational Site 13888, Providence, Rhode Island
  - Teva Investigational Site 13871, Charleston, South Carolina
  - Teva Investigational Site 13889, Charleston, South Carolina
  - Teva Investigational Site 13853, Spartanburg, South Carolina
  - Teva Investigational Site 14671, Summerville, South Carolina
  - Teva Investigational Site 13898, Baytown, Texas
  - Teva Investigational Site 14673, Boerne, Texas
  - Teva Investigational Site 13867, El Paso, Texas
  - Teva Investigational Site 13902, Killeen, Texas
  - Teva Investigational Site 13846, Live Oak, Texas
  - Teva Investigational Site 13878, San Antonio, Texas
  - Teva Investigational Site 14672, San Antonio, Texas
  - Teva Investigational Site 13917, San Antonio, Texas
  - Teva Investigational Site 13845, Waco, Texas
  - Teva Investigational Site 13850, Richmond, Virginia
  - Teva Investigational Site 13915, Bellingham, Washington
- Georgia (8):
  - Teva Investigational Site 81041, Kutaisi
  - Teva Investigational Site 81047, Tbilisi
  - Teva Investigational Site 81046, Tbilisi
  - Teva Investigational Site 81044, Tbilisi
  - Teva Investigational Site 81040, Tbilisi
  - Teva Investigational Site 81045, Tbilisi
  - Teva Investigational Site 81042, Tbilisi
  - Teva Investigational Site 81043, Tbilisi
- Hungary (10):
  - Teva Investigational Site 51277, Budapest
  - Teva Investigational Site 51278, Budapest
  - Teva Investigational Site 51272, Budapest
  - Teva Investigational Site 51279, Debrecen
  - Teva Investigational Site 51271, Dombóvár
  - Teva Investigational Site 51269, Győr
  - Teva Investigational Site 51274, Kaposvár
  - Teva Investigational Site 51270, Miskolc
  - Teva Investigational Site 51276, Szeged
  - Teva Investigational Site 51273, Szigetvár
- Russia (9):
  - Teva Investigational Site 50444, Moscow
  - Teva Investigational Site 50446, Perm
  - Teva Investigational Site 50442, Saint Petersburg
  - Teva Investigational Site 50447, Saint Petersburg
  - Teva Investigational Site 50441, Saint Petersburg
  - Teva Investigational Site 50448, Saint Petersburg
  - Teva Investigational Site 50445, Saint Petersburg
  - Teva Investigational Site 50443, Saint Petersburg
  - Teva Investigational Site 50440, Tomsk
- Ukraine (14):
  - Teva Investigational Site 58261, Chernivtsi
  - Teva Investigational Site 58262, Dnipropetrovsk
  - Teva Investigational Site 58269, Ivano-Frankivsk
  - Teva Investigational Site 58270, Kharkiv
  - Teva Investigational Site 58265, Kryvyi Rih
  - Teva Investigational Site 58271, Kyiv
  - Teva Investigational Site 58268, Kyiv
  - Teva Investigational Site 58264, Kyiv
  - Teva Investigational Site 58260, Lviv
  - Teva Investigational Site 58259, Odesa
  - Teva Investigational Site 58272, Odesa
  - Teva Investigational Site 58263, Vinnytsia
  - Teva Investigational Site 58267, Zaporizhzhia
  - Teva Investigational Site 58266, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 841 participants with persistent asthma were randomized in a 1:1:1:1 ratio to receive Fp MDPI 25 mcg, Fp MDPI 50 mcg, FS MDPI 50/12.5 mcg, or placebo MDPI. Randomization was stratified by previous therapy (inhaled corticosteroid [ICS] or non-corticosteroid [NCS]).
Groups:
- Fp MDPI 25 mcg BID: Participants received 1 inhalation of 25 micrograms (mcg) fluticasone propionate (Fp) via MDPI twice daily (BID) (total daily dose: 50 mcg) for 12 weeks.
Period: Overall Study
Arm/Group | Placebo MDPI | Fp MDPI 25 mcg BID | Fp MDPI 50 mcg BID | FS MDPI 50/12.5 mcg BID
Started | 209 | 211 | 210 | 211
Received at Least 1 Dose of Study Drug (Safety analysis set) | 209 | 211 | 208 | 211
Completed | 202 | 206 | 203 | 205
Not Completed | 7 | 5 | 7 | 6
Not completed — Other than specified | 1 | 1 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 3
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by parent/guardian | 6 | 3 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all randomized participants.
Groups:
- Placebo MDPI: Participants received matching placebo via MDPI for 12 weeks.
- Fp MDPI 25 mcg BID: Participants received 1 inhalation of 25 mcg fluticasone propionate via MDPI BID (total daily dose: 50 mcg) for 12 weeks.
- FS MDPI 50/12.5 mcg BID: Participants received 1 inhalation of 50/12.5 mcg fluticasone propionate/salmeterol via MDPI BID (total daily dose: 100/25 mcg) for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo MDPI | Fp MDPI 25 mcg BID | Fp MDPI 50 mcg BID | FS MDPI 50/12.5 mcg BID | Total
Number analyzed (Participants) | 209 | 211 | 210 | 211 | 841
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.5 (1.98) | 8.7 (1.83) | 8.5 (1.94) | 8.4 (2.05) | 8.5 (1.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 74 | 80 | 91 | 324
  Male | 130 | 137 | 130 | 120 | 517
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 172 | 168 | 171 | 172 | 683
  Black or African American | 33 | 41 | 32 | 29 | 135
  Asian | 1 | 0 | 2 | 3 | 6
  American Indian or Alaska Native | 0 | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Other | 2 | 1 | 3 | 7 | 13
At-Home Baseline Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: percent predicted of FEV1] — FEV1 is the volume of air exhaled in the first second of a forced expiration as measured by spirometer. Baseline trough morning percent predicted FEV1 was defined as the average value of recorded (nonmissing) morning assessments 5 out of the last 7 days prior to randomization. Population: Here, 'Number analyzed' signifies participants evaluable for this parameter.
  percent predicted of FEV1
    number analyzed (Participants) | 209 | 211 | 209 | 211 | 840
    (all) | 68.8 (9.70) | 69.6 (9.68) | 69.6 (9.47) | 69.9 (9.15) | 69.5 (9.49)
In-Clinic Baseline Percent Predicted FEV1 [Mean (Standard Deviation); unit: percent predicted of FEV1] — FEV1 is the volume of air exhaled in the first second of a forced expiration as measured by spirometer. The baseline 1-hour trough morning percent predicted FEV1 was defined as the predose trough morning percent predicted FEV1 measurement at the randomization visit (Baseline [Day 1]) at the investigational center. 'Number of participants analyzed' for this parameter are 209, 211, 209, and 211 for each arm respectively. Population: Here, 'Number analyzed' signifies participants evaluable for this parameter.
  percent predicted of FEV1
    number analyzed (Participants) | 209 | 211 | 209 | 211 | 840
    (all) | 74.9 (14.58) | 73.0 (13.43) | 72.9 (13.00) | 74.1 (15.02) | 73.7 (14.03)

OUTCOME MEASURES:

1. Primary Outcome: For FS MDPI Versus Fp MDPI: Change From Baseline in 1-Hour Postdose Percent Predicted Morning Forced Expiratory Volume in 1 Second (FEV1) at Week 12
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer. The baseline 1-hour trough morning percent predicted FEV1 was defined as the predose trough morning percent predicted FEV1 measurement at the randomization visit (Baseline [Day 1]) at the investigational center. The IMP dose was administered right after the predose FEV1 measurement (within a 10 minute window). Participant then performed 1-hour (±10 minutes) postdose lung function assessments on Week 12 at the investigational center.
Time Frame: Baseline, Week 12
Population: ITT analysis set included all randomized participants. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure. Missing data was imputed using MNAR methodology for prematurely discontinue participants or MAR for completers with implausible data.
Measure: Least Squares Mean (Standard Error); unit: percent predicted of FEV1
Arm/Group | Fp MDPI 25 mcg BID | Fp MDPI 50 mcg BID | FS MDPI 50/12.5 mcg BID
Number analyzed (Participants) | 211 | 209 | 211
percent predicted of FEV1 | 16.8 (1.32) | 16.4 (1.32) | 18.2 (1.29)
Statistical Analysis 1: Comparison: Fp MDPI 50 mcg BID vs FS MDPI 50/12.5 mcg BID; Analysis was performed using an ANCOVA model with effects due to baseline trough morning percent predicted FEV1, sex, age, (pooled) investigational center, previous therapy (ICS or NCS), and IMP treatment group; Test type: Superiority; p = 0.285, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = 1.9, 95% CI 2-sided [-1.6 to 5.3]

2. Primary Outcome: For Fp MDPI Versus Placebo: Change From Baseline in Weekly Average of the Percent Predicted Trough Morning FEV1 at Week 12
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer. Baseline trough morning percent predicted FEV1 was defined as the average value of recorded (nonmissing) morning assessments 5 out of the last 7 days prior to randomization. The first day before randomization consisted of the electronic patient diary entry at home on the morning of the randomization visit (Baseline [Day 1]) and the first day postrandomization consisted of the electronic patient diary entry at home on the morning of the day after the randomization visit (Baseline [Day 1]). For postdose weekly average of trough morning percent predicted FEV1 measurements, the values were the averages based on the available data for that week. The averages were calculated as the sum of morning FEV1 values divided by the number of nonmissing assessments.
Time Frame: Baseline, Week 12
Population: ITT analysis set included all randomized participants. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure. Missing data was imputed using missing not at random (MNAR) methodology for prematurely discontinue participants or missing at random (MAR) for completers with implausible data.
Measure: Least Squares Mean (Standard Error); unit: percent predicted of FEV1
Arm/Group | Placebo MDPI | Fp MDPI 25 mcg BID | Fp MDPI 50 mcg BID
Number analyzed (Participants) | 209 | 211 | 209
percent predicted of FEV1 | 7.3 (1.10) | 13.3 (1.09) | 14.2 (1.10)
Statistical Analysis 1: Comparison: Placebo MDPI vs Fp MDPI 25 mcg BID; Analysis was performed using an analysis of covariance (ANCOVA) model with effects due to baseline trough morning percent predicted FEV1, sex, age, (pooled) investigational center, previous therapy (inhaled corticosteroid [ICS] or noncorticosteroid [NCS]), and investigational medicinal product (IMP) treatment group; Test type: Superiority; p < 0.001, ANCOVA — Threshold for significance at 0.05 level; Least square (LS) mean difference = 6.0, 95% CI 2-sided [3.2 to 8.8]
Statistical Analysis 2: Comparison: Placebo MDPI vs Fp MDPI 50 mcg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = 7.0, 95% CI 2-sided [4.1 to 9.8]

3. Secondary Outcome: Change From Baseline in the Weekly Average of Daily Trough Morning (Predose and Pre-Rescue Bronchodilator) Peak Expiratory Flow (PEF) Over the 12 Week Treatment Period
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. Morning PEF was determined in the morning, before administration of IMP or rescue medications. Baseline trough morning PEF was defined as the average value of recorded (nonmissing) morning assessments 5 out of the last 7 days prior to randomization. The first day before randomization consisted of the electronic patient diary entry at home on the morning of the randomization visit (Baseline [Day 1]) and the first day postrandomization consisted of the electronic patient diary entry at home on the morning of the day after the randomization visit (Baseline [Day 1]). For postdose weekly average of trough morning PEF measurements, the values were the averages based on the available data for that week. The averages were calculated as the sum of morning PEF values divided by the number of nonmissing assessments.
Time Frame: Baseline, Week 1 to 12
Population: ITT analysis set included all randomized participants. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Placebo MDPI | Fp MDPI 25 mcg BID | Fp MDPI 50 mcg BID | FS MDPI 50/12.5 mcg BID
Number analyzed (Participants) | 208 | 210 | 208 | 211
liters/minute | 12.3 (2.65) | 28.9 (2.62) | 26.3 (2.64) | 32.0 (2.61)

4. Secondary Outcome: Change From Baseline in the Weekly Average of Total Daily (24 Hour) Use of Albuterol/Salbutamol Inhalation Aerosol (Number of Inhalations) Over Weeks 1 Through 12
Description: Participants recorded the number of inhalations of rescue medication (albuterol/salbutamol HFA MDI) each morning and evening in the electronic patient diary. An entry of 0 inhalations indicated no rescue medication was needed. To calculate the total daily use of albuterol/salbutamol inhalation aerosol (number of inhalations), the electronic patient diary entry on randomization visit (Baseline [Day 1]) was defined as the first day of analysis. The weekly average of the total daily inhalations was the average based on the available data for that week. The average was calculated as the sum of total daily inhalations over the 7 days for each analysis week divided by the number of nonmissing assessments. LS mean and standard error (SE) were obtained using mixed model for repeated measures (MMRM).
Time Frame: Baseline, Week 1 to 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: inhalations
Arm/Group | Placebo MDPI | Fp MDPI 25 mcg BID | Fp MDPI 50 mcg BID | FS MDPI 50/12.5 mcg BID
Number analyzed (Participants) | 208 | 210 | 209 | 211
inhalations | -0.2 (0.05) | -0.4 (0.05) | -0.5 (0.05) | -0.4 (0.05)

5. Secondary Outcome: Change From Baseline in the Weekly Average of the Total Daily Asthma Symptom Score Over Weeks 1 Through 12
Description: Asthma symptom scores were recorded in the patient diary. Each participant assessed the symptoms of cough, wheeze, shortness of breath, and chest tightness and entered a single score that was inclusive of all symptoms. Daytime Symptom Score (determined in the evening) ranged from 0=No symptoms during the day to 5=Symptoms so severe that I could not go to work or perform normal daily activities. Nighttime Symptom Score (determined in the morning) ranged from 0=No symptoms during the night to 4=Symptoms so severe that I did not sleep at all. The total daily asthma symptom score was the average of the daytime and nighttime scores. The total daily asthma symptom score ranged from 0 - 9 with 0=no symptoms during the day or night and 9=severe symptoms both day and night. The weekly average was calculated as the sum of total daily asthma symptom scores over the 7 days for each analysis week divided by the number of nonmissing assessments. LS mean and SE were obtained using MMRM.
Time Frame: Baseline, Week 1 to 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo MDPI | Fp MDPI 25 mcg BID | Fp MDPI 50 mcg BID | FS MDPI 50/12.5 mcg BID
Number analyzed (Participants) | 208 | 210 | 209 | 211
units on a scale | -0.1 (0.02) | -0.2 (0.02) | -0.2 (0.02) | -0.2 (0.02)

6. Secondary Outcome: Change From Baseline in Asthma Control (Measured by Childhood Asthma Control Test [C-ACT] Score) Over the 12 Week Treatment Period
Description: C-ACT was a simple, participant-completed tool used for the assessment of overall asthma control. The first 4 items of the test were completed by the participant, while the last 3 items were completed by the participant's parents/legal guardians/caregivers. A total sum score based upon responses to all items was calculated to provide an overall measure of asthma control. The derived C-ACT score ranging from 0 to 27. These scores spanned the continuum of poor control of asthma (score ≤5) to complete control of asthma (score ≥25), with a cut off score of 19 indicating participants with poorly controlled asthma. LS mean and SE were obtained using MMRM.
Time Frame: Baseline, Week 1 to 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo MDPI | Fp MDPI 25 mcg BID | Fp MDPI 50 mcg BID | FS MDPI 50/12.5 mcg BID
Number analyzed (Participants) | 204 | 208 | 205 | 209
units on a scale | 4.5 (0.21) | 5.1 (0.21) | 5.5 (0.21) | 5.4 (0.21)

7. Secondary Outcome: Time to First Onset of Effect
Description: The time to first onset of effect, defined as the first decrease from baseline in daily rescue medication use, was calculated based on the number of inhalations of rescue medication (albuterol/salbutamol hydrofluoroalkane metered-dose inhaler [HFA MDI] [90 mcg ex actuator] or equivalent) recorded by the participant each morning and evening in the patient diary built into the handheld device.
Time Frame: Baseline up to Week 12
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo MDPI | Fp MDPI 25 mcg BID | Fp MDPI 50 mcg BID | FS MDPI 50/12.5 mcg BID
Number analyzed (Participants) | 208 | 210 | 208 | 211
days | 20.0 [5.0 to NA] — Due to smaller number of participants with an event, upper limit of 95% confidence interval (CI) could not be calculated. | NA [3.0 to NA] — Due to smaller number of participants with an event, median and upper limit of 95% CI could not be calculated. | 2.0 [2.0 to 2.0] | 6.0 [2.0 to NA] — Due to smaller number of participants with an event, upper limit of 95% CI could not be calculated.

8. Secondary Outcome: Percentage of Participants Who Discontinued From Investigational Medicinal Product (IMP) for Asthma Exacerbation During the 12 Week Treatment Period
Time Frame: Baseline up to Week 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo MDPI | Fp MDPI 25 mcg BID | Fp MDPI 50 mcg BID | FS MDPI 50/12.5 mcg BID
Number analyzed (Participants) | 208 | 210 | 208 | 211
percentage of participants | 6 | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: Baseline up to Week 13
Description: Safety analysis set included all randomized participants who received at least 1 dose of IMP.
Arm/Group | Placebo MDPI | Fp MDPI 25 mcg BID | Fp MDPI 50 mcg BID | FS MDPI 50/12.5 mcg BID
All-Cause Mortality (participants affected / at risk) | 0/209 | 0/211 | 0/208 | 0/211
Serious Adverse Events (participants affected / at risk) | 1/209 | 2/211 | 1/208 | 4/211
Other Adverse Events (participants affected / at risk) | 11/209 | 8/211 | 11/208 | 9/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo MDPI (N=209) | Fp MDPI 25 mcg BID (N=211) | Fp MDPI 50 mcg BID (N=208) | FS MDPI 50/12.5 mcg BID (N=211)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disruptive mood dysregulation disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo MDPI (N=209) | Fp MDPI 25 mcg BID (N=211) | Fp MDPI 50 mcg BID (N=208) | FS MDPI 50/12.5 mcg BID (N=211)
Nasopharyngitis (Infections and infestations) | 11 (12) | 8 (9) | 11 (11) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT02980133/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT02980133/SAP_001.pdf